CLINICAL TRIAL: NCT00572559
Title: A Randomized, Open Label, Multi-Center Clinical Trial, Comparing Microbiologic Response To Linezolid And Vancomycin In Ventilator-Associated Pneumonia (VAP) Due To Methicillin Resistant Staphylococcus Aureus (MRSA)
Brief Title: Microbiologic Response With Linezolid And Vancomycin In Ventilator-Associated Pneumonia Due To Methicillin Resistant Staphylococcus Aureus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 766-INF-0026-126; A5951069
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2010-06

CONDITIONS: Pneumonia, Ventilator-Associated
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Vancomycin; Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Vancomycin
- 2 (Experimental)
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: Vancomycin — 1 gram IV every 12 hours for 7 to 14 days
  Arms: 1
Drug: Linezolid — 600 mg every 12 hours (intravenously [IV] for a minimum of the first 4 days followed by a switch to oral if tolerated by patient) for a total duration of 7 to 14 days
  Arms: 2

SUMMARY:
Ventilator-associated pneumonia (VAP) is a commonplace complication of intensive care patients ventilated for longer than 48 hours. Methicillin-resistant Staphylococcus aureus (MRSA) is the cause of late onset VAP in up to about 30% of cases in US hospitals. Ineffective treatment of MRSA VAP clearly leads to prolonged mechanical ventilation and is probably associated with higher mortality. The purpose of this protocol is to directly compare linezolid and vancomycin specifically for MRSA VAP.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have or be suspected of having a ventilator-associated pneumonia (VAP) due to MRSA.
* Patient must be hospitalized for at least 5 days, must be ventilator-dependent ≥ 48 hours prior to screen/baseline, and anticipated to remain on the ventilator for 72 hours after enrollment so follow-up BAL can be performed.
* Clinical picture compatible with pneumonia (acquired during ventilation)
* Chest X Ray at baseline/screen or within 24 hours of initiation of therapy must be consistent with diagnosis of pneumonia

Exclusion Criteria:

* Hypersensitivity to linezolid, vancomycin, or one of the excipients in any of these drug formulations.
* Infections due to gram-positive organisms known to be resistant to either of the study drugs.
* Any antibiotic used in the treatment of MRSA, such as vancomycin, TMP/SMX, rifampin, or linezolid, for more than 48 hours prior to patient's enrollment into the study.
* Patients with neutropenia, AIDS, lymphoma or anticipated chemotherapy.
* Patients who have long-term tracheostomy (for more than 60 days). Acute tracheostomy patients are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2002-11; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
To assess early microbiologic response in patients with VAP due to MRSA based on semi-quantitative culture of bronchoscopic bronchoalveolar lavage (BAL) in patients treated with linezolid vs vancomycin. | 72-96 hours

SECONDARY OUTCOMES:
To compare duration of mechanical ventilation | 0000
To compare post treatment tracheal colonization | FU: 14 days after EOT +/- 2 days
To identify clinical correlates of infection based on microbiologic sampling as determined by original and modified CPIS (Clinical Pulmonary Infection Score) | EOT: Day 14; FU: 14 days after EOT +/- 2 days
To compare the microbiological cure based on BAL specimens with the traditional criteria for microbiologic cure | 72-96 hours
To compare mortality at End Of Treatment (EOT) and Follow up (FU); To compare clinical outcome at EOT and FU | EOT: Day 14; FU: 14 days after EOT +/- 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (26):
- United States (25):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Palm Springs, California
  - Pfizer Investigational Site, Rancho Mirage, California
  - Pfizer Investigational Site, Redlands, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, Norwalk, Connecticut
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Augusta, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, North East Atlanta, Georgia
  - Pfizer Investigational Site, ‘Ewa Beach, Hawaii
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Peoria, Illinois
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, Cortland Manor, New York
  - Pfizer Investigational Site, Jamaica, New York
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Morgantown, West Virginia
- Pfizer Investigational Site, San Juan, Puerto Rico

REFERENCES:
- [Derived] Wunderink RG, Mendelson MH, Somero MS, Fabian TC, May AK, Bhattacharyya H, Leeper KV Jr, Solomkin JS. Early microbiological response to linezolid vs vancomycin in ventilator-associated pneumonia due to methicillin-resistant Staphylococcus aureus. Chest. 2008 Dec;134(6):1200-1207. doi: 10.1378/chest.08-0011. Epub 2008 Aug 21. PMID 18719064